CLINICAL TRIAL: NCT02951156
Title: PHASE 1B/PHASE 3 MULTICENTER STUDY OF AVELUMAB (MSB0010718C) IN COMBINATION REGIMENS THAT INCLUDE AN IMMUNE AGONIST, EPIGENETIC MODULATOR, CD20 ANTAGONIST AND/OR CONVENTIONAL CHEMOTHERAPY IN PATIENTS WITH RELAPSED OR REFRACTORY DIFFUSE LARGE B-CELL LYMPHOMA (DLBCL) JAVELIN DLBCL
Brief Title: Avelumab In Combination Regimens That Include An Immune Agonist, Epigenetic Modulator, CD20 Antagonist and/or Conventional Chemotherapy in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL)
Acronym: Javelin DLBCL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to closure of study arms following futility analysis and difficulty in enrolling participants due to evolving treatment landscape
Sponsor: Pfizer (Industry)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991011; 2016-002904-15 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2016-11-01 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — avelumab; utomilumab; Rituximab; Azacitidine; Bendamustine Hydrochloride; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1b Arm A (Experimental): avelumab/utomilumab/rituximab
  Interventions: Biological: Avelumab; Biological: Utomilumab; Biological: Rituximab
- Phase 1b Arm B (Experimental): avelumab/utomilumab/azacitidine
  Interventions: Biological: Avelumab; Biological: Utomilumab; Other: Azacitidine
- Phase 1b Arm C (Experimental): avelumab/rituximab/bendamustine
  Interventions: Biological: Avelumab; Biological: Rituximab; Drug: Bendamustine
- Phase 3 Arm D (selected from Phase 1b) (Experimental): Selected regimen from Phase 1b component which may be i) avelumab/utomilumab/rituximab OR ii) avelumab/rituximab/azacitidine OR iii) avelumab/rituximab/bendamustine
  Interventions: Biological: Avelumab; Biological: Utomilumab; Biological: Rituximab; Other: Azacitidine; Drug: Bendamustine
- Phase 3 Arm E (Active Comparator): Investigator's Choice of either rituximab/bendamustine or rituximab/gemcitabine/oxaliplatin
  Interventions: Biological: Rituximab; Drug: Bendamustine; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Avelumab — Investigational fully human anti-PD-L1 monoclonal antibody
  Other Names: MSB0010718C
  Arms: Phase 1b Arm A; Phase 1b Arm B; Phase 1b Arm C; Phase 3 Arm D (selected from Phase 1b)
Biological: Utomilumab — Investigational, fully human IgG2 CD 137/4-1BB agonist
  Other Names: PF-05082566
  Arms: Phase 1b Arm A; Phase 1b Arm B; Phase 3 Arm D (selected from Phase 1b)
Biological: Rituximab — CD20-directed cytolytic antibody
  Other Names: Rituxan
  Arms: Phase 1b Arm A; Phase 1b Arm C; Phase 3 Arm D (selected from Phase 1b); Phase 3 Arm E
Other: Azacitidine — Antimetabolite antineoplastic agent and demethylation agent.
  Other Names: Vidaza
  Arms: Phase 1b Arm B; Phase 3 Arm D (selected from Phase 1b)
Drug: Bendamustine — Alkylating drug
  Other Names: Treanda
  Arms: Phase 1b Arm C; Phase 3 Arm D (selected from Phase 1b); Phase 3 Arm E
Drug: Gemcitabine — Nucleoside analogue
  Other Names: Gemzar
  Arms: Phase 3 Arm E
Drug: Oxaliplatin — Platinum-based drug
  Other Names: Eloxatin
  Arms: Phase 3 Arm E

SUMMARY:
Study B9991011 is a multi-center, international, randomized, open label, 2 component (Phase 1b followed by Phase 3), parallel-arm study of avelumab in combination with various agents for the treatment of Relapsed/Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL).

DETAILED DESCRIPTION:
The target study population of this Phase 1b/3 registrational study is patients with R/R DLBCL who have completed at least 2 (but not more than 4) lines of prior rituximab-containing multi-agent chemotherapy, and/or in whom autologous stem cell transplant (ASCT) has failed, or who are not candidates for ASCT or who are not eligible for intensive chemotherapy. Patients who are ineligible for intensive second line chemotherapy must have received at least one prior rituximab-containing combination chemotherapy regimen. The study will assess the safety, efficacy, pharmacokinetics (PK), immunogenicity of the 3 avelumab-based combination regimens tested, and collect patient reported outcome (PRO) data.

ELIGIBILITY:
Key Inclusion Criteria:

-Any of the following as defined by the WHO, 2016 lymphoid neoplasm classifications and histologically confirmed:

* Diffuse large B-cell lymphoma (DLBCL), Not Otherwise Specified (NOS): Germinal center B-cell type (GCB), Activated B-cell type (ABC)
* High-grade B-cell lymphoma (HGBCL) NOS
* HGBCL with MYC and BCL2 and/or BCL6 rearrangements
* T-cell histocyte-rich large B-cell lymphoma
* EBV+ DLBCL, NOS
* HHV8+ DLBCL, NOS

Relapsed or refractory disease following at least 2 lines (and a maximum of 4 lines) of prior rituximab containing multi-agent chemotherapy which may include an autologous stem cell transplantation unless patients are not considered suitable for intensive second-line chemotherapy or autologous stem cell transplantation. Patients who are ineligible for intensive second line chemotherapy,must have received at least one prior rituximab-containing combination chemotherapy regimen. Patients who are ineligible for intensive second line chemotherapy, must have received at least one prior rituximab-containing combination chemotherapy regimen.

* Baseline measurable disease with at least 1 bi dimensional lesion with longest diameter (LDi) >1.5cm on CT scan which is FDG avid on PET scan.
* A biopsy (archived or Screening/recent) will be collected at Screening.
* At least 18years of age (or ≥20 years in Japan).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.

Key Exclusion Criteria:

* Active central nervous system (CNS) lymphoma.
* Prior organ transplantation including prior allogeneic SCT.
* Prior therapy with an anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab, tremelimumab or any other antibody, or drug specifically targeting T cell co stimulatory or immune checkpoint pathways).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (9):
  - City of Hope, Duarte, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Norton Diagnostic Center - Dupont, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Parexel International, Billerica, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - North Shore Hematology Oncology Associates, East Setauket, New York
- Australia (4):
  - St. George Hospital, Kogarah, New South Wales
  - Monash Health, Clayton, Victoria
  - Cancer Clinical Trials Centre, Austin Health, Level 4, Heidelberg, Victoria
  - Genesis Care, Heidelberg, Victoria
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Italy (2):
  - Farmacia Studi Clinici, Rozzano, MI
  - Istituto Clinico Humanitas, Rozzano, MI
- Poland (5):
  - Malopolskie Centrum Medyczne S.C., Krakow, Lesser Poland Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej im. Sw. Jana z Dukli, Lublin, Lublin Voivodeship
  - Nzoz McD Voxel Osrodek Pet-Tk-Nmr, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. Sw. Jana z Dukli Oddzial Hematologiczny, Lublin
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej Zamosc Sp. z o.o., Zamość
- South Korea (2):
  - Samsung Medical Center Clinical Trial Pharmacy, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital San Pedro de Alcantara, Cáceres
  - Centro de Investigación Medicina Especializada Sanitaria (CIMES), Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - The Christie Pathology Partnership, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hawkes EA, Phillips T, Budde LE, Santoro A, Saba NS, Roncolato F, Gregory GP, Verhoef G, Offner F, Quero C, Radford J, Giannopoulos K, Stevens D, Thall A, Huang B, Laird AD, Sandner R, Ansell SM. Avelumab in Combination Regimens for Relapsed/Refractory DLBCL: Results from the Phase Ib JAVELIN DLBCL Study. Target Oncol. 2021 Nov;16(6):761-771. doi: 10.1007/s11523-021-00849-8. Epub 2021 Oct 23. PMID 34687398
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) after completion of at least 2 and not more than 4 lines of rituximab-containing multi-agent chemotherapy (prior to this study), and/or in whom autologous stem cell transplant (ASCT) has failed, or who were not candidates for ASCT or who were not eligible for intensive chemotherapy.
Pre-assignment Details: This study was planned to be conducted into two phases: Phase 1b and Phase 3. Phase 3 of the study was never conducted due to early termination of study because of Phase 1b enrollment closure.
Groups:
- Avelumab+Rituximab+Utomilumab: Avelumab 10 milligram per kilogram (mg/kg) intravenous (IV) infusion was administered every 2 weeks on Day 2 and Day 16 of Cycles 1 and 2, if well tolerated then continued on Day 1 and Day 15 in Cycle 3 and all subsequent cycles, until the participant no longer received clinical benefit. Rituximab 375 milligram per meter square (mg/m^2) IV infusion was administered on Day 1 of each treatment cycle (maximum of 8 cycles), along with fixed dose of 100 mg IV infusion of utomilumab on Day 2 of each treatment cycle in Cycles 1 and 2. If the dose of utomilumab was well tolerated, then it was administered on Day 1 of Cycle 3 and all subsequent cycles until the participant no longer received clinical benefit. The duration of each treatment cycle was 28 days.
- Avelumab+Azacitidine+Utomilumab: Avelumab 10 mg/kg IV infusion was administered every 2 weeks on Day 2 and Day 16 of Cycles 1 and 2, if well tolerated then continued on Day 1 and Day 15 in Cycle 3 and all subsequent cycles, until the participant no longer received clinical benefit. Azacitidine 40 mg/m^2 subcutaneous (SC) dose was administered on Days 1 to 5 of each treatment cycle until the participant no longer received clinical benefit, along with fixed dose of 100 mg IV infusion of utomilumab on Day 2 of each treatment cycle in Cycles 1 and 2. If the dose of utomilumab was well tolerated, then it was administered on Day 1 of Cycle 3 and all subsequent cycles until the participant no longer received clinical benefit. The duration of each treatment cycle was 28 days.
- Avelumab+Bendamustine+Rituximab: Avelumab 10 mg/kg IV infusion was administered every 2 weeks on Day 2 and Day 16 of Cycles 1 and 2, if well tolerated then continued on Day 1 and Day 15 in Cycle 3 and all subsequent cycles, until the participant no longer received clinical benefit. Rituximab 375 mg/m^2 IV infusion was administered on Day 1 of each treatment cycle (maximum of 8 cycles), along with 90 mg/m^2 IV infusion of bendamustine on Day 2 and Day 3 of each treatment cycle in Cycles 1 and 2. If the dose of bendamustine was well tolerated, then it was administered on Day 1 and Day 2 in Cycle 3 and all subsequent cycles for a maximum of 6 cycles. The duration of each treatment cycle was 28 days.
Period: Overall Study
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Started | 9 | 9 | 11
Completed | 0 | 0 | 1
Not Completed | 9 | 9 | 10
Not completed — Death | 3 | 8 | 5
Not completed — Progressive disease | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 1
Not completed — Other | 5 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Avelumab+Rituximab+Utomilumab: Avelumab 10 mg/kg IV infusion was administered every 2 weeks on Day 2 and Day 16 of Cycles 1 and 2, if well tolerated then continued on Day 1 and Day 15 in Cycle 3 and all subsequent cycles, until the participant no longer received clinical benefit. Rituximab 375 mg/m^2 IV infusion was administered on Day 1 of each treatment cycle (maximum of 8 cycles), along with fixed dose of 100 mg IV infusion of utomilumab on Day 2 of each treatment cycle in Cycles 1 and 2. If the dose of utomilumab was well tolerated, then it was administered on Day 1 of Cycle 3 and all subsequent cycles until the participant no longer received clinical benefit. The duration of each treatment cycle was 28 days.
- Avelumab+Azacitidine+Utomilumab: Avelumab 10 mg/kg IV infusion was administered every 2 weeks on Day 2 and Day 16 of Cycles 1 and 2, if well tolerated then continued on Day 1 and Day 15 in Cycle 3 and all subsequent cycles, until the participant no longer received clinical benefit. Azacitidine 40 mg/m^2 SC dose was administered on Days 1 to 5 of each treatment cycle until the participant no longer received clinical benefit, along with fixed dose of 100 mg IV infusion of utomilumab on Day 2 of each treatment cycle in Cycles 1 and 2. If the dose of utomilumab was well tolerated, then it was administered on Day 1 of Cycle 3 and all subsequent cycles until the participant no longer received clinical benefit. The duration of each treatment cycle was 28 days.
- Total: Total of all reporting groups
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab | Total
Number analyzed (Participants) | 9 | 9 | 11 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5 | 10
  >=65 years | 7 | 6 | 6 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 9 | 6 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 11 | 26
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 8 | 8 | 11 | 27
  Race: Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: AEs occurring in first 4 weeks of treatment,attributable to 1 of study drugs. Hematology:1)Grade 4 neutropenia,2)Grade >=3 febrile neutropenia with single temperature of >38.3 degrees Celsius (C)/sustained temperature of >=38.0 degrees C for more than 1 hour with/without associated sepsis,3)Grade >=3 neutropenic infection,4)Grade 4 thrombocytopenia/Grade 3 thrombocytopenia with clinically significant bleeding,5)Grade 4 anemia 6)Any grade >=3 non-hematology toxicity except:transient Grade 3 flu like symptoms/fever controlled with standard medical management;transient Grade 3 fatigue,localized skin reactions/headache that resolves to Grade <=1;Grade 3 nausea,vomiting/diarrhea resolved to Grade <=1 in ˂72 hours after initiation of adequate medical management;Grade 3 skin toxicity resolved to Grade <=1 in ˂7 days;tumor flare;Single laboratory values that are out of normal range,that have no clinical correlate and resolve to Grade <=1 within 7 days with adequate medical management.
Time Frame: Day 1 Cycle 1 up to 4 Weeks
Population: DLT evaluable set included all participants who were randomized in the study and received at least 1 dose of study medication and either experienced DLT during the first cycle, or completed the primary DLT observation period of 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 7 | 5 | 10
Participants | 1 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR) as Assessed by Investigator Per Lugano Response Classification Criteria
Description: ORR was defined as percentage of participants with complete response (CR) or partial response (PR), as assessed by investigator per lugano response classification criteria. CR was defined as a score of 1 (no uptake above background), 2 (uptake less than or equal to [<=] mediastinum), or 3 (uptake less than [<] mediastinum but <=liver) with or without a residual mass on PET 5-point scale (5-PS), for lymph nodes and extralymphatic sites; no new lesions; no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. PR was defined as >=50% decrease in SPD of up to six of the largest dominant lymph nodes, no increase in size of other nodes, liver, or spleen volume, a >=50% decrease in sum of products of diameters (SPD) of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease.
Time Frame: Randomization until date of PD, start of new anticancer therapy, discontinuation from study or death due to any cause, whichever occurred first (maximum up to 36 months)
Population: Full analysis set population included all participants who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 9 | 9 | 11
Percentage of participants | 11.1 [0.3 to 48.2] | 0 [0.0 to 33.6] | 27.3 [6.0 to 61.0]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Greater Than or Equal to (>=) Grade 3, As Per National Cancer Institute Common Terminology Criteria For Adverse Events (NCI-CTCAE), Version 4.03
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03,severity was graded as Grade 1:asymptomatic/mild symptoms,clinical/diagnostic observations only, intervention not indicated; Grade 2:moderate, minimal, local/noninvasive intervention indicated,limiting age-appropriate instrumental activities of daily life (ADL); Grade 3:severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4:life-threatening consequence, urgent intervention indicated; Grade 5:death related to AE. TEAE was defined as events which occurred during on-treatment period beginning with first dose of study treatment through minimum (30 days + last dose of study treatment or start of new anti-cancer drug therapy). In this outcome measure participant with any TEAE of Grade 3 or above are reported.
Time Frame: From first dose of study treatment up to at least 30 days after the last dose of study treatment or initiation of new anti-cancer therapy (up to 36 months)
Population: Safety analysis set population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
Participants | 4 | 7 | 10

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities As Per National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Laboratory parameters included hematological and biochemistry: Hematological parameters included: anemia, haemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and white blood cells decreased. Biochemistry parameters included alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, cholesterol high, creatine kinase(cpk) increased, creatinine increased, gamma glutamyl transferase(ggt) increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypertriglyceridemia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase increased,serum amylase increased.Test abnormalities were graded by NCI CTCAE version 4.03 as Grade 1=mild; Grade 2=moderate; Grade 3/Grade 4=severe/life-threatening. Number of participants with abnormalities of any grade were reported.
Time Frame: as for outcome 3
Population: Safety analysis set population included all participants who received at least 1 dose of study drug. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
Participants
  Anemia: number analyzed (Participants) | 8 | 8 | 10
  Anemia | 6 | 8 | 10
  Hemoglobin increased: number analyzed (Participants) | 8 | 8 | 10
  Hemoglobin increased | 0 | 0 | 0
  Lymphocyte count decreased: number analyzed (Participants) | 7 | 8 | 10
  Lymphocyte count decreased | 4 | 7 | 9
  Lymphocyte count increased: number analyzed (Participants) | 7 | 8 | 10
  Lymphocyte count increased | 0 | 0 | 0
  Neutrophil count decreased: number analyzed (Participants) | 8 | 8 | 10
  Neutrophil count decreased | 2 | 2 | 9
  Platelet count decreased: number analyzed (Participants) | 8 | 8 | 10
  Platelet count decreased | 4 | 3 | 8
  White blood cell decreased: number analyzed (Participants) | 7 | 8 | 10
  White blood cell decreased | 1 | 4 | 8
  Alanine aminotransferase increased: number analyzed (Participants) | 7 | 8 | 10
  Alanine aminotransferase increased | 2 | 5 | 2
  Alkaline phosphatase increased: number analyzed (Participants) | 7 | 8 | 10
  Alkaline phosphatase increased | 3 | 4 | 6
  Aspartate aminotransferase increased: number analyzed (Participants) | 7 | 8 | 9
  Aspartate aminotransferase increased | 3 | 6 | 3
  Blood bilirubin increased: number analyzed (Participants) | 7 | 8 | 10
  Blood bilirubin increased | 0 | 3 | 3
  Cholesterol high: number analyzed (Participants) | 7 | 7 | 10
  Cholesterol high | 2 | 3 | 3
  Cpk increased: number analyzed (Participants) | 7 | 7 | 10
  Cpk increased | 2 | 1 | 2
  Creatinine increased: number analyzed (Participants) | 7 | 8 | 10
  Creatinine increased | 6 | 6 | 10
  GGT increased: number analyzed (Participants) | 7 | 7 | 10
  GGT increased | 3 | 4 | 6
  Hypercalcemia: number analyzed (Participants) | 7 | 8 | 10
  Hypercalcemia | 0 | 3 | 2
  Hyperglycemia: number analyzed (Participants) | 7 | 8 | 10
  Hyperglycemia | 3 | 1 | 2
  Hyperkalemia: number analyzed (Participants) | 8 | 8 | 10
  Hyperkalemia | 0 | 0 | 2
  Hypermagnesemia: number analyzed (Participants) | 7 | 8 | 10
  Hypermagnesemia | 1 | 1 | 1
  Hypernatremia: number analyzed (Participants) | 7 | 8 | 10
  Hypernatremia | 0 | 0 | 1
  Hypertriglyceridemia: number analyzed (Participants) | 7 | 6 | 10
  Hypertriglyceridemia | 3 | 3 | 7
  Hypoalbuminemia: number analyzed (Participants) | 7 | 8 | 10
  Hypoalbuminemia | 3 | 4 | 6
  Hypocalcemia: number analyzed (Participants) | 7 | 8 | 10
  Hypocalcemia | 1 | 0 | 2
  Hypoglycemia: number analyzed (Participants) | 7 | 8 | 10
  Hypoglycemia | 0 | 0 | 1
  Hypokalemia: number analyzed (Participants) | 8 | 8 | 10
  Hypokalemia | 1 | 1 | 4
  Hypomagnesemia: number analyzed (Participants) | 7 | 8 | 10
  Hypomagnesemia | 0 | 0 | 4
  Hyponatremia: number analyzed (Participants) | 7 | 8 | 10
  Hyponatremia | 0 | 1 | 3
  Hypophosphatemia: number analyzed (Participants) | 7 | 7 | 10
  Hypophosphatemia | 1 | 0 | 5
  Lipase increased: number analyzed (Participants) | 7 | 7 | 10
  Lipase increased | 1 | 2 | 3
  Serum amylase increased: number analyzed (Participants) | 7 | 7 | 10
  Serum amylase increased | 2 | 1 | 3

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities included: 1) QT interval, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF): increase from baseline greater than (>) 30 millisecond (ms) or 60 ms; absolute value >450 ms, >480 ms and >500 ms; 2) heart rate (HR): absolute value <=50 beats per minute (bpm) and decrease from baseline >=20 bpm; absolute value >=120 bpm and increase from baseline >=20 bpm; 3) PR interval: absolute value >=220 ms and increase from baseline >=20 ms; 4) QRS interval: absolute value >=120 ms.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
Participants
  QT: Increase from baseline >30 ms | 4 | 4 | 4
  QT: Increase from baseline >60 ms | 1 | 3 | 2
  QT: >450 ms | 2 | 2 | 2
  QT: >480 ms | 0 | 1 | 1
  QT: >500 ms | 0 | 0 | 0
  QTcB: Increase from baseline >30 ms: number analyzed (Participants) | 7 | 9 | 10
  QTcB: Increase from baseline >30 ms | 1 | 3 | 4
  QTcB: Increase from baseline >60 ms: number analyzed (Participants) | 7 | 9 | 10
  QTcB: Increase from baseline >60 ms | 1 | 1 | 0
  QTcB: >450 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcB: >450 ms | 4 | 5 | 9
  QTcB: >480 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcB: >480 ms | 2 | 3 | 4
  QTcB: >500 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcB: >500 ms | 1 | 2 | 1
  QTcF: Increase from baseline >30 ms: number analyzed (Participants) | 7 | 9 | 10
  QTcF: Increase from baseline >30 ms | 1 | 3 | 3
  QTcF: Increase from baseline >60 ms: number analyzed (Participants) | 7 | 9 | 10
  QTcF: Increase from baseline >60 ms | 0 | 2 | 0
  QTcF: >450 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcF: >450 ms | 4 | 3 | 6
  QTcF: >480 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcF: >480 ms | 0 | 2 | 0
  QTcF: >500 ms: number analyzed (Participants) | 7 | 9 | 11
  QTcF: >500 ms | 0 | 2 | 0
  Heart rate: <=50 bpm and decrease from baseline >=20 bpm: number analyzed (Participants) | 7 | 9 | 10
  Heart rate: <=50 bpm and decrease from baseline >=20 bpm | 0 | 1 | 0
  Heart rate: >=120 bpm and increase from baseline >=20 bpm: number analyzed (Participants) | 7 | 9 | 10
  Heart rate: >=120 bpm and increase from baseline >=20 bpm | 0 | 0 | 1
  PR: >=220 ms and increase from baseline >=20 ms: number analyzed (Participants) | 8 | 8 | 11
  PR: >=220 ms and increase from baseline >=20 ms | 0 | 0 | 0
  QRS: >=120 ms | 1 | 1 | 2

6. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator Per Lugano Response Classification Criteria
Description: Investigator assessed DOR: was defined for participants with OR as time from first documentation of OR to time of first documentation of disease progression/death due to any cause, whichever occurred first. CR: score of 1(no uptake above background),2(uptake <=mediastinum),or 3(uptake <mediastinum but <=liver) with or without a residual mass on PET 5-PS,for lymph nodes extralymphatic sites;no new lesions;no evidence of FDG-avid disease in bone marrow. PR: >=50% decrease in SPD of up to 6 of largest dominant lymph nodes,no increase in size of other nodes,liver,spleen volume,>=50% decrease in SPD of hepatic splenic nodules,absence of other organ involvement,no new sites of disease. PD: appearance of new lesion more than 1.5 cm in any axis,at least a 50% increase from nadir in SPD/longest diameter of previous lesion/node. Data was censored on date of last adequate tumor assessment in participants with no event,started new anti-cancer therapy/had 2 or more missing assessments.
Time Frame: First response (CR or PR) to date of PD, start of new anti-cancer therapy, discontinuation from the study, censoring date or death due to any cause, whichever occurred first (maximum up to 36 months)
Population: Participants who were randomized and achieved an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 1 | 0 | 3
Months | 1.81 [1.81 to 1.81] |  | NA [NA to NA] — Median and full range could not be calculated as all 3 participants who achieved OR were not observed to have PD or death on study

7. Secondary Outcome: Time to Tumor Response (TTR) as Assessed by Investigator Per Lugano Response Classification Criteria
Description: TTR was defined for participants who achieved objective response as time from randomization to first documentation of objective tumor response (CR or PR) that was subsequently confirmed. CR was defined as a score of 1 (no uptake above background), 2 (uptake <= mediastinum), or 3 (uptake <mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow. PR was defined as >=50% decrease in SPD of up to six of the largest dominant lymph nodes, no increase in size of other nodes, liver, or spleen volume, a >=50% decrease in SPD of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease.
Time Frame: From the date of randomization to the first documentation of objective response (CR or PR) (maximum up to 36 months)
Population: Participants who were randomized and achieved an objective response.
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 1 | 0 | 3
Months | 1.8 [1.8 to 1.8] |  | 1.9 [1.7 to 2.6]

8. Secondary Outcome: Disease Control Rate as Assessed by the Investigator Per Lugano Response Classification Criteria
Description: Disease control rate was defined as percentage of participants with disease control. Disease Control (DC) was defined as the best overall response of CR, PR, or stable disease (SD). CR: score of 1 (no uptake above background), 2 (uptake <= mediastinum), or 3 (uptake less than <mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow. PR: >=50% decrease in SPD of up to six of the largest dominant lymph nodes, no increase in size of other nodes, liver, or spleen volume, a >=50% decrease in SPD of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease. SD: <50% decrease in SDP of up to 6 dominant, measurable nodes and extranodal sites; no criteria for progressive disease met. To qualify as a best overall response of SD, at least one SD assessment must be observed >=6 weeks after start date and before disease progression.
Time Frame: From the date of randomization to the first documentation of PD, study discontinuation, start of new anti-cancer therapy or death due to any cause, whichever occurred first (maximum up to 36 months)
Population: Full analysis set population included all participants who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 9 | 9 | 11
Percentage of participants | 22.2 [2.8 to 60.0] | 0 [0 to 33.6] | 36.4 [10.9 to 69.2]

9. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator Per Lugano Response Classification Criteria
Description: Investigator assessed PFS was defined as time (in months) from date of randomization to the first documentation of disease progression or death (due to any cause), whichever occurred first. PFS data was censored on the date of the last adequate tumor assessment for participants who had no an event (PD or death), for participants who start a new anti-cancer therapy prior to an event or for participants with an event after 2 or more missing or inadequate post-baseline tumor assessment. Participants without an adequate baseline or post-baseline tumor assessment were censored on the date of randomization unless death occurred on or before the time of the second planned tumor assessment in which case the death was considered as an event.
Time Frame: From the date of randomization to progression of disease, study discontinuation, censoring date or death due to any cause, whichever occurred first (up to 36 months)
Population: Full analysis set population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 9 | 9 | 11
Months | 1.8 [0.6 to 3.5] | 1.5 [0.3 to 1.8] | 2.7 [1.3 to NA] — Due to small number of participants who had events, upper limit of 95% CI was not estimable.

10. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From the date of randomization to discontinuation from the study or death, whichever occurred first (maximum up to 36 months)
Population: Full analysis set population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 9 | 9 | 11
Months | 14.8 [0.9 to NA] — Due to small number of participants who had events, upper limit of 95% CI was not estimable. | 4.0 [0.3 to 11.3] | 5.2 [1.3 to NA] — Due to small number of participants who had events, upper limit of 95% CI was not estimable.

11. Secondary Outcome: Concentration Verses Time Summary of Avelumab
Time Frame: 1 hour Post dose Day 2 Cycle 1, 144 hour Post dose Day 8 of Cycle 1, 0 hour Post dose Day 16 of Cycle 1, Day 1 of Cycle 4 and Cycle 6
Population: Avelumab pharmacokinetic concentration analysis set included all participants who received at least 1 dose of study drug and who had at least 1 post-dose concentration measurement above the lower limit of quantitation for avelumab. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
microgram per milliliter (mcg/mL)
  Cycle 1 Day 2: number analyzed (Participants) | 7 | 7 | 10
  Cycle 1 Day 2 | 183.29 (83.809) | 198.43 (29.387) | 193.30 (29.702)
  Cycle 1 Day 8: number analyzed (Participants) | 8 | 8 | 10
  Cycle 1 Day 8 | 75.14 (21.357) | 68.44 (18.553) | 65.33 (17.913)
  Cycle 1 Day 16: number analyzed (Participants) | 7 | 4 | 9
  Cycle 1 Day 16 | 25.33 (13.197) | 26.53 (9.237) | 19.36 (7.810)
  Cycle 4 Day 1: number analyzed (Participants) | 2 | 1 | 4
  Cycle 4 Day 1 | 25.00 (4.667) | 62.00 (NA) — Due to single participant with data available for this outcome measure at this time point, Standard Deviation was not estimable. | 120.88 (165.187)
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 4
  Cycle 6 Day 1 |  | 7.57 (NA) — Due to single participant with data available for this outcome measure at this time point, Standard Deviation was not estimable. | 39.43 (18.327)

12. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Avelumab by Never and Ever Positive Status
Description: ADA never-positive was defined as no positive ADA results at any time point. ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Baseline: 2 hours pre-dose of first dose of avelumab, Post baseline: post first dose up to up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Avelumab immunogenicity analysis set included participants who had at least 1 ADA sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
Participants
  Baseline: ADA ever-positive | 0 | 0 | 1
  Baseline: ADA never-positive | 8 | 9 | 10
  Post Baseline: ADA ever-positive | 0 | 0 | 0
  Post Baseline: ADA never-positive | 8 | 9 | 11

13. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Rituximab by Never and Ever Positive Status
Description: as for outcome 12
Time Frame: From the date of first study treatment up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Rituximab immunogenicity analysis set included participants who had at least 1 ADA sample collected for rituximab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 11
Participants
  ADA ever-positive | 0 | 0
  ADA never-positive | 8 | 11

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Utomilumab by Never and Ever Positive Status
Description: as for outcome 12
Time Frame: From the date of first study treatment up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Utomilumab immunogenicity analysis set included participants who had at least 1 ADA sample collected for utomilumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab
Number analyzed (Participants) | 8 | 9
Participants
  ADA ever-positive | 1 | 2
  ADA never-positive | 7 | 7

15. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Avelumab by Never and Ever Positive Status
Description: nAb never-positive was defined as no positive nAb results at any time point and nAb ever-positive was defined as at least one positive nAb result at any time point.
Time Frame: From the date of first study treatment up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Data for this outcome measure was not collected since there was no participants with post-baseline ADA ever positive sample for avelumab.
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Rituximab by Never and Ever Positive Status
Description: as for outcome 15
Time Frame: From the date of first study treatment up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Data for this this outcome measure was not collected since there was no participant with rituximab ADA ever positive sample.
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Utomilumab by Never and Ever Positive Status
Description: as for outcome 15
Time Frame: From the date of first study treatment up to 30 Days after the end of treatment (maximum up to 36 months)
Population: Utomilumab immunogenicity analysis set included participants from the safety analysis set who had at least one ADA/nAb sample collected for utomilumab. Here, 'overall number of participants analyzed' signifies number of participants who were ADA positive and whose samples were further analyzed for nAb.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab
Number analyzed (Participants) | 1 | 2
Participants
  nAb ever-positive | 0 | 0
  nAb never-positive | 1 | 2

18. Secondary Outcome: Programmed Death Receptor-1 Ligand-1 (PD-L1) Biomarker Expression in Tumor and Immune Cells as Assessed by Immunohistochemistry (IHC) at Baseline
Description: Percentage of Tumor and Immune Cells as Assessed by Immunohistochemistry at Baseline.
Time Frame: Screening (prior to first dose of study treatment)
Population: Full analysis set population included all participants who were randomized in the study. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Percentage of cells staining positive
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 6 | 8 | 6
Percentage of cells staining positive
  Tumor Cells (membrane) | 0 [0 to 5] | 0.5 [0.0 to 10.0] | 0 [0 to 30]
  Immune Cells | 7.5 [0.0 to 30.0] | 7.5 [0.0 to 70.0] | 17.5 [0.0 to 50.0]

19. Secondary Outcome: Number of Participants With Minimal Residual Disease Burden (MRD) Positive, Negative and Not Evaluable (NE) Status
Description: Number of participants with MRD positive, negative and not evaluable status were reported in this outcome measure.
Time Frame: Baseline, Day 1 of Cycle 3, 6, 9, 12 and 18
Population: Safety analysis set population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
Number analyzed (Participants) | 8 | 9 | 11
Participants
  Baseline: Positive | 3 | 1 | 3
  Baseline: Negative | 0 | 0 | 2
  Baseline: NE | 5 | 8 | 6
  Cycle 3 Day 1: Positive | 3 | 1 | 1
  Cycle 3 Day 1: Negative | 0 | 0 | 3
  Cycle 3 Day 1: NE | 2 | 1 | 1
  Cycle 6 Day 1: Positive | 0 | 1 | 0
  Cycle 6 Day 1: Negative | 0 | 0 | 2
  Cycle 6 Day 1: NE | 0 | 0 | 2
  Cycle 9 Day 1: Positive | 0 | 0 | 0
  Cycle 9 Day 1: Negative | 0 | 0 | 1
  Cycle 9 Day 1: NE | 0 | 0 | 2
  Cycle 12 Day 1: Positive | 0 | 0 | 0
  Cycle 12 Day 1: Negative | 0 | 0 | 1
  Cycle 12 Day 1: NE | 0 | 0 | 2
  Cycle 18 Day 1: Positive | 0 | 0 | 0
  Cycle 18 Day 1: Negative | 0 | 0 | 0
  Cycle 18 Day 1: NE | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to follow up (36 months)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set population included all participants who received at least 1 dose of study drug.
Arm/Group | Avelumab+Rituximab+Utomilumab | Avelumab+Azacitidine+Utomilumab | Avelumab+Bendamustine+Rituximab
All-Cause Mortality (participants affected / at risk) | 4/8 | 8/9 | 6/11
Serious Adverse Events (participants affected / at risk) | 3/8 | 6/9 | 7/11
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab+Rituximab+Utomilumab (N=8) | Avelumab+Azacitidine+Utomilumab (N=9) | Avelumab+Bendamustine+Rituximab (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab+Rituximab+Utomilumab (N=8) | Avelumab+Azacitidine+Utomilumab (N=9) | Avelumab+Bendamustine+Rituximab (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Asthenia (General disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium (Investigations) | 0 | 0 | 1
Blood chloride increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 3 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2
Generalised oedema (General disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lipase decreased (Investigations) | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 3
Malaise (General disorders) | 0 | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 5
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Primary hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Data for Phase 3 outcome measures were not collected as study was terminated early and phase 3 was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02951156/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02951156/SAP_001.pdf